CLINICAL TRIAL: NCT04790695
Title: Single Patient Protocol for an NRG1 Fusion Positive Metastatic Pancreatic Cancer Patient Using Seribantumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOHCC-OLIP-01
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — seribantumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Seribantumab (Experimental): For the induction phase: Seribantumab 3,000 mg IV weekly for 12 weeks then Maintenance Phase: Seribantumab 3,000 mg IV infusion once every 2 weeks, initiating approximately 14 days after completion of induction phase. Dose or schedule may be adjusted at the discretion of the treating physician.
  Interventions: Drug: Seribantumab

INTERVENTIONS:
Drug: Seribantumab — For the induction phase: Seribantumab 3,000 mg IV weekly for 12 weeks then Maintenance Phase: Seribantumab 3,000 mg IV infusion once every 2 weeks, initiating approximately 14 days after completion of induction phase. Dose or schedule may be adjusted at the discretion of the treating physician.

SUMMARY:
NRG1 gene fusions are extremely rare across solid tumours (estimate 0.3-0.5%). However, it is felt to be an actionable and potentially major growth pathway for those tumours that harbour this gene rearrangement. Tumours that harbour NRG1 fusions are driven by HER3 overactivation. Seribantumab is a mono-clonal antibody against HER3, it binds HER3 and inhibits NRG1-dependent activation and HER2 dimerization.

ELIGIBILITY:
Inclusion Criteria:

* Serious, life-threatening condition

  * Not eligible for, or exhausted all other treatment options or causing significant toxicity
  * No other way to access treatment

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No